CLINICAL TRIAL: NCT03886649
Title: Copanlisib in Combination With Venetoclax in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma. A Multicenter Phase Ib Trial With Two Expansion Cohorts
Brief Title: Copanlisib in Combination With Venetoclax in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Funding
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 66/18
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Relapsed or refractory B-cell non-Hodgkin lymphoma; Copanlisib; Venetoclax; Non-Hodgkin lymphoma; Splenic marginal zone lymphoma; Extranodal marginal zone lymphoma of mucosa-associated lymphoid tissue (MALT lymphoma); Nodal marginal zone lymphoma; Follicular lymphoma; Diffuse large B-cell lymphoma (DLBCL), NOS
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Lymphoma, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Dendritic Cell Sarcoma, Interdigitating | interventions — copanlisib; venetoclax

STUDY DESIGN:
Intervention Model Description: In the dose escalation phase, relapsed/refractory B-cell NHL patients are included. In the dose expansion phase, patients with MZL (Marginal zone lymphoma) and FL (Follicular lymphoma) will be treated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copanlisib + Venetoclax (Experimental): Phase Ib -> dose escalation with 2 expansion cohorts
  Interventions: Drug: Copanlisib; Drug: Venetoclax

INTERVENTIONS:
Drug: Copanlisib — Duration of IMP administration: a maximum of twelve 28-day cycles of the combination treatment. Copanlisib will be administered i.v. on days 1, 8, and 15 of each cycle. The only dose level 1 (DL1) is 60 mg copanlisib.
Drug: Venetoclax — Duration of IMP administration: a maximum of twelve 28-day cycles of the combination treatment. Copanlisib will be administered i.v. on days 1, 8, and 15 of each cycle. The starting dose is dose level 1 (DL1): 600 mg venetoclax.

SUMMARY:
A significant number of patients with non-Hodgkin lymphoma (NHL) are not cured with available treatments and will eventually relapse. Those patients might not be able to tolerate more bone marrow toxicity, limiting their treatment options. Preclinical in vitro studies have demonstrated a synergism of venetoclax and copanlisib in different lymphomas. This may represent a safe and effective therapy for patients who relapsed or did not respond to standard therapy.

The primary objective of this phase I trial is to establish the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of copanlisib in combination with venetoclax in patients with relapsed or refractory B-cell NHL.

DETAILED DESCRIPTION:
There are many different types of NHL. A lot of progress has been made over the last years in the management of NHL, and while some can be cured with available treatments, for others new treatments are necessary. A significant number of patients that cannot be cured with the available treatments will eventually relapse.

Dysregulation of apoptosis via overexpression of the antiapoptotic BCL-2 protein is paramount for several subtypes of NHL. On the other hand, PI3K is a central pathway in the pathogenesis of lymphoma, and PI3K signaling is critical for the proliferation and survival of malignant cells such as follicular lymphoma (FL), marginal zone lymphoma (MZL), and others.

The combination of copanlisib (PI3K inhibitor) and venetoclax (BLC-2 inhibitor) is interesting given their known single agent activity in B-cell NHL and their synergy observed in B-cell NHL preclinical models. The pharmacologic inhibition of PI3K by copanlisib has translated into significant clinical activity in different lymphoma subtypes. Venetoclax has proven successful in CLL and the first results in NHL are encouraging. Both compounds are currently in other combination studies in SLL/CLL and NHL but there are currently no clinical trials studying this particular combination.

There is a need to further improve approaches in the relapsed/refractory setting of patients with NHL in need of systemic therapy and this combination may provide an opportunity for an active and well-tolerated regimen that does not present the short and long-term toxicities of chemotherapy.

The phase Ib study here proposed will evaluate the safety, tolerability and preliminary antitumor activity of the novel combination of copanlisib with venetoclax, two drugs with single agent activity across different lymphoma subtypes in the dose escalation and in two small cohorts of patients with FL and MZL in the expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration and prior to any trial specific procedures.
* Histologically confirmed B-cell NHL lymphoma as per WHO classification for the escalation phase. FL or MZL for the expansion phase.
* Patients with relapsed or refractory disease who have failed previous treatment (including chemotherapy plus anti CD20) for whom no effective standard treatment is available or refused by the patient.
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence.
* > 1 two-dimensionally measurable nodal lesion in CT, PET/CT scan (preferable) or MRI, according to Cheson et al, 2014.
* Tumor tissue (formalin fixed paraffin embedded (FFPE) slides/rolls) is available for the mandatory translational research.
* Age ≥ 18 years.
* WHO performance status 0-1
* Adequate bone marrow function:

  1. Absolute neutrophil count (ANC) >1.5 × 109/l (1 × 109/l if due to bone marrow involvement by lymphoma). Patient must not have received any hematologic growth factor within 14 days prior to registration.
  2. Platelet count >100 ×109/l (75 ×109/l if due to bone marrow involvement by lymphoma)
* Adequate hepatic function:

  1. total bilirubin ≤ 1.5 × ULN (except for patients with Gilbert's disease ≤ 3.0 × ULN),
  2. AST and ALT ≤ 2.5 × ULN, or ≤ 5 × ULN under the assumption that abnormal values are tumor related.
* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 50 ml/min/1.73 m2 (according to CKD-EPI formula)
* Adequate cardiac function: Left ventricular Ejection Fraction (LVEF) ≥ 50% as determined by echocardiography (ECHO).
* Adequate coagulation function: INR ≤ 1.5 × ULN (the ULN for INR is defined with the value 1.2 for all sites, in case no ULN is documented in the lab certificates/sheets), aPTT ≤ 1.5 × ULN.
* Women of childbearing potential (not surgically sterile or exceeding 2 years after the onset of menopause) must use highly effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 3 months after the last dose of investigational drug. A negative pregnancy test before inclusion into the trial is required for all women of childbearing potential.
* Men agree not to donate sperm or to father a child during trial treatment and until 3 months after the last dose of investigational drug.
* Patient is able and willing to swallow trial drug as whole tablet.

Exclusion Criteria:

* Patients with CLL/SLL.
* Patients that require ramp-up of venetoclax, including MCL. Other histologies will be discussed with the coordinating investigator (CI).
* Presence or history of CNS disease (either CNS lymphoma or lymphomatous meningeosis). Primary CNS disease.
* Prior treatment with venetoclax, copanlisib or any other bcl-2 inhibitors or PIK3 inhibitors.
* Prior allogeneic stem cell transplant (SCT), or autologous transplant less than 3 months prior to registration.
* Concomitant or recent treatment with any other experimental drug (enrollment in another clinical trial.
* Treatment with any anti-lymphoma therapies within 21 days prior to registration - except for local radiation therapy for palliative treatment of symptoms.
* Not resolved grade ≥ 2 (per NCI CTCAE v5.0 toxicity (other than alopecia) from prior therapy at registration.
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV; (see Appendix 4), unstable or new onset angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation.
* Uncontrolled hypertension (sustained systolic blood pressure >150 mmHg and or diastolic >90 mmHg) despite optimal medical management (per investigator's assessment).
* Proteinuria of ≥ CTCAE grade 3 as assessed by a 24h total urine protein quantification or on a random urine sample, estimated by urine protein to creatinine ratio > 3.5.
* HbA1c > 8.5%.
* Lipase ≥ 1.5 x ULN.
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to registration.
* Major surgery within 1 month prior to registration.
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment. All patients must be screened for HIV up to 28 days prior to study drug start using a blood test for HIV according to local regulations. All patients must be screened for hepatitis up to 28 days prior to study drug start using the routine hepatitis virus laboratory panel. Patients positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.
* Active CMV infection. Patients who are CMV PCR positive at baseline will be excluded.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Concomitant or prior use of immunosuppressive medication within 28 days before registration, with the exceptions of intranasal and inhaled corticosteroids, or systemic corticosteroids which must not exceed 10 mg/day of prednisone or a dose equivalent corticosteroid).
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Concomitant anticoagulation treatment with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon), factor Xa inhibitors (e.g. rivaroxaban, apixaban), direct thrombin inhibitors (e.g. dabigatran) or platelet inhibitors/antiplatelet agents. Exception: Aspirin (up to 300 mg/day) is allowed.
* Concomitant treatment with strong CYP3A inducers or inhibitors (see http://medicine.iupui.edu/ and the FDA database of drug interactions. Concomitant treatment with moderate inhibitors or inducers during the DLT period.
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information.
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s).
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) during the first cycle of treatment | day 28 of the first cycle
  Dose-limiting toxicity (DLT) is defined as any of the adverse events (AEs) which:
  * occurs during cycle 1 of the trial treatment (defined as the DLT monitoring period), and
  * is considered by the investigator or the sponsor to be at least possibly related to at least one of the drugs given in the combination trial treatment venetoclax+copanlisib.

SECONDARY OUTCOMES:
Adverse events (AEs) | at 12 months
Complete response (CR) at 6 months and 12 months | at 6 months and 12 months
Overall response (OR) at 6 months and 12 months | at 6 months and 12 months
OR based on best response | at 12 months
Progression-free survival (PFS) at 12 months | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Stathis, MD, Study Chair — IOSI, Ospedale San Giovanni, Bellinzona; Emanuele Zucca, Study Chair — IOSI, Ospedale San Giovanni, Bellinzona
Locations (6):
- Switzerland (6):
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich